CLINICAL TRIAL: NCT03579927
Title: Immunotherapy With Ex Vivo-Expanded Cord Blood-Derived CAR-NK Cells Combined With High-Dose Chemotherapy and Autologous Stem Cell Transplantation for B-Cell Lymphoma
Brief Title: CAR.CD19-CD28-zeta-2A-iCasp9-IL15-Transduced Cord Blood NK Cells, High-Dose Chemotherapy, and Stem Cell Transplant in Treating Participants With B-cell Lymphoma
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of Funding
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0295; NCI-2018-01111 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0295 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2018-06-25; First posted 2018-07-09 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: CD19 Positive; Mantle Cell Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Filgrastim; Granulocyte Colony-Stimulating Factor; Melphalan; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CAR transduced CB-NK cells, chemotherapy, ASCT) (Experimental): Participants receive rituximab IV over 3 hours on days -14 and -8, carmustine IV over 2 hours on day -13, etoposide IV over 3 hours BID on days -12 to -9, cytarabine IV over 1 hour BID on days -12 to -9, melphalan IV over 30 minutes on day -8, CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced CB-NK cells IV over 1 hour on day -5. Participants undergo ASCT on day 0. Beginning day 0, participants receive filgrastim SC QD until evidence of an ANC of 0.5 x 10^9/L per 3 consecutive days.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Biological: Filgrastim; Drug: Melphalan; Biological: Rituximab; Biological: Umbilical Cord Blood-derived Natural Killer Cells

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo ASCT
  Other Names: Autologous Hematopoietic Cell Transplantation; autologous stem cell transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Biological: Filgrastim — Given SC
  Other Names: FILGRASTIM, LICENSE HOLDER UNSPECIFIED; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine nitrogen mustard; Sarcoclorin; Sarkolysin; WR-19813
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
Biological: Umbilical Cord Blood-derived Natural Killer Cells — Given CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced CB-NK cells IV
  Other Names: Cord Blood NK Cells; Umbilical Cord Blood-derived NK Cells

SUMMARY:
This phase I/II trial studies the side effects and best dose of chimeric antigen receptor (CAR).CD19-CD28-zeta-2A-iCasp9-IL15-transduced cord blood NK cells when given together with high-dose chemotherapy and stem cell transplant and to see how well they work in treating participants with B-cell lymphoma. Cord blood-derived CAR-NK cells may react against the B-cell lymphoma cells in the body, which may help to control the disease. Giving chemotherapy before a stem cell transplant may help kill any cancer cells that are in the body and helps make room in the patient's bone marrow for new blood-forming cells (stem cells) to grow. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the safety and relative efficacy of CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced cord blood natural killer (CB-NK) cells in patients with B cell non-Hodgkin lymphoma (NHL) undergoing high dose chemotherapy and autologous stem cell transplantation.

SECONDARY OBJECTIVES:

I. To estimate the relapse-free survival (RFS). II. To estimate the overall survival (OS). III. To quantify the persistence of infused CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced CB-NK cells in the recipient.

OUTLINE: This is a phase I, dose-escalation study of CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced CB-NK cells followed by a phase II study.

Participants receive rituximab intravenously (IV) over 3 hours on days -14 and -8, carmustine IV over 2 hours on day -13, etoposide IV over 3 hours twice daily (BID) on days -12 to -9, cytarabine IV over 1 hour BID on days -12 to -9, melphalan IV over 30 minutes on day -8, CAR.CD19-CD28-zeta-2A-iCasp9-IL15-transduced CB-NK cells IV over 1 hour on day -5. Participants undergo autologous stem cell transplantation (ASCT) on day 0. Beginning day 0, participants receive filgrastim subcutaneously (SC) once daily (QD) until evidence of an absolute neutrophil count (ANC) of 0.5 x 10^9/L per 3 consecutive days.

After completion of study treatment, participants are followed for up to 15 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70.
2. Patients with B-cell lymphoma who are candidates to autologous stem-cell transplantation, including: 1. Primary refractory or relapsed diffuse large B-cell lymphoma in response to salvage treatment. 2. Primary refractory or relapsed follicular lymphoma or other indolent B-cell histology in response to salvage treatment. 3. Chemosensitive mantle-cell lymphoma in first or later line of treatment. 4. Patients with B cell lymphoma (all CD19+ NHL) with progressive or refractory disease who would otherwise not be candidates for autologous stem cell transplantation.
3. Adequate organ function: Renal: Creatinine clearance (as estimated by Cockcroft Gault) >/= 60 cc/min. Hepatic: ALT/AST </= 2.5 x ULN or </= 5 x ULN if documented liver metastases, Total bilirubin </= 1.5 mg/dL, except in subjects with Gilbert's Syndrome in whom total bilirubin must be </= 3.0 mg/dL. Cardiac: Cardiac ejection fraction >/= 50%, no evidence of pericardial effusion as determined by an ECHO, and no clinically significant ECG findings. Pulmonary: No clinically significant pleural effusion, Baseline oxygen saturation > 92% on room air.
4. Patients must have a cord blood unit available which is matched with the patient at 4, 5, or 6/6 HLA class I (serological) and II (molecular) antigens.
5. Availability of autologous peripheral blood stem cell graft, containing at least 6.0 x 10^6 CD34+ cells/kg.
6. Performance status < 2 (ECOG).
7. Negative Beta HCG in woman with child-bearing potential.
8. All participants who are able to have children must practice effective birth control while on study. Acceptable forms of birth control for female patients include: hormonal birth control, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence, for the length of the study. If the participant is a female and becomes pregnant or suspects pregnancy, she must immediately notify her doctor. If the participant becomes pregnant during this study, she will be taken off this study. Men who are able to have children must use effective birth control while on the study. If the male participant fathers a child or suspects that he has fathered a child while on the study, he must immediately notify his doctor.
9. Signed consent to long-term follow-up protocol PA17-0483.

Exclusion Criteria:

1. Primary CNS lymphoma.
2. Grade >/= 3 non-hematologic toxicity from prior therapy that has not resolved to </= G1.
3. Prior whole brain irradiation.
4. Active hepatitis B, either active carrier (HBsAg +) or viremic (HBV DNA >/= 10,000 copies/mL, or >/= 2,000 IU/mL).
5. Evidence of either cirrhosis or stage 3-4 liver fibrosis in patients with chronic hepatitis C or positive hepatitis C serology.
6. Active infection requiring parenteral antibiotics.
7. HIV infection.
8. Radiation therapy in the month prior to enroll.
9. Presence of fungal, bacterial, viral, or other infection requiring IV antimicrobials for management. Note: Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment.
10. Concomitant use of other investigational agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events defined as graft failure, grade 3, 4 graft versus host disease, grade 3,4 cytokine release syndrome, grade 3, 4, neuro-toxicity, or death from any cause | Up to 30 days within natural killer (NK) cell infusion
  Frequencies of toxicity will be summarized by dose. The relationships between toxicity and efficacy as functions of dose and other covariates will be assessed by fitting Bayesian regression models.
Complete response (CR) or partial response (PR) | At day 30 post NK cell infusion
  Efficacy is defined as the patient being alive and in CR or PR at day 30 post NK cell infusion. Frequencies of efficacy will be summarized by dose. The relationships between toxicity and efficacy as functions of dose and other covariates will be assessed by fitting Bayesian regression models.

SECONDARY OUTCOMES:
Progression-free survival (PFS) time | At day 100
  Unadjusted distributions of the time-to-event outcome PFS will be estimated using the method of Kaplan and Meier. The relationship of PFS to prognostic covariates and NK cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Overall survival (OS) time | At day 100
  Unadjusted distributions of the time-to-event outcome OS will be estimated using the method of Kaplan and Meier. The relationship of OS to prognostic covariates and NK cell dose level will be evaluated by Bayesian piecewise exponential survival regression.
Response status | 16 weeks
  Participants have a bone marrow aspiration and/or biopsy to check the status of the disease.
Number of chimeric antigen receptor (CAR) NK cells in blood by flow cytometry | Up to 16 weeks post CAR NK cell infusion
  The number of CAR NK cells in blood by flow cytometry will be measured on days 3, 7, 14, 21, and at 4 weeks, 8 weeks, 12 weeks, and 16 weeks post CAR NK cell infusion. In addition to preliminary graphical analysis to assess possible patterns over time Bayesian longitudinal regression using a generalized Poisson regression model for the count at each time point as a function of patient baseline covariates, and random latent patient effects to induce within-patient correlation among each patient's vector of CAR NK cell counts.

CONTACTS AND LOCATIONS:
Overall Officials: Katy Rezvani, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org